CLINICAL TRIAL: NCT03714191
Title: Using Rapid Cycle Randomized Controlled Trials to Study a Tobacco Cessation Best Practice Advisory.
Brief Title: Optimizing the Tobacco Cessation Clinical Decision Support Tool.
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-Tobacco Cessation
Record Dates: First submitted 2018-10-04; First posted 2018-10-22 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Social Control, Formal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Improved outcomes
  Interventions: Other: Patient Outcomes
- Regulatory reminder
  Interventions: Other: Regulatory
- Billing and documentation
  Interventions: Other: Billing documentation

INTERVENTIONS:
Other: Patient Outcomes — The intervention includes different versions of the BPA design and message.
  Groups: Improved outcomes
Other: Billing documentation — The intervention includes different versions of the BPA design and message.
  Groups: Billing and documentation
Other: Regulatory — The intervention includes different versions of the BPA design and message.
  Groups: Regulatory reminder

SUMMARY:
The existing tobacco cessation best practice advisory (BPA) fires for providers (physicians, residents, fellows, midwives, nurse practitioners, physician assistants) during outpatient encounters when a patient is identified as a current tobacco user in the Social History section of their chart. The BPA was designed to help facilitate tobacco cessation interventions; it is part of the The Centers for Medicare & Medicaid Services (CMS) Quality Payment Program (QPP). The purpose of the project is to optimize this BPA utilization and improve patient outcomes by comparing multiple versions of the tobacco cessation BPA.

ELIGIBILITY:
Inclusion Criteria:

* All providers of patients at NYU Langone Health (including NYU Winthrop) who are identified as currents smokers, as documented in the social history of their patient chart, and are eligible to receive the best practice advisory for tobacco cessation.

Exclusion Criteria:

* non smokers

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All providers of patients at NYU Langone Health (including NYU Winthrop) who are identified as currents smokers, as documented in the social history of their patient chart, and are eligible to receive the best practice advisory for tobacco cessation.
Sampling Method: Probability Sample
Enrollment: 54417 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Alert acceptance rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Austrian J, Mendoza F, Szerencsy A, Fenelon L, Horwitz LI, Jones S, Kuznetsova M, Mann DM. Applying A/B Testing to Clinical Decision Support: Rapid Randomized Controlled Trials. J Med Internet Res. 2021 Apr 9;23(4):e16651. doi: 10.2196/16651. PMID 33835035